CLINICAL TRIAL: NCT04461223
Title: Evaluation of Myocardial Injury After Anthracycline Chemotherapy in Osteosarcoma Patients Using CMR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-523
Record Dates: First submitted 2020-06-28; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2019-12

CONDITIONS: Cardiotoxicity; Osteosarcoma; Myocardial Injury; Chemotherapy Induced Systolic Dysfunction; Doxorubicin Induced Cardiomyopathy
Keywords: Osteosarcoma; CMR; T1 mapping, T2 mapping, T2* mapping, LGE, ECV
MeSH Terms: conditions — Cardiotoxicity; Osteosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: contrast-enhanced cardiac magnetic resonance imaging(MAGNETOM Aera 1.5T) — CMR T1 mapping, T2mapping, T2* mapping, LGE, ECV
  Other Names: CMR

SUMMARY:
using a contrast-enhanced (CE) cardiac magnetic resonance imaging(CMR) which included the measurement of T1 mapping, T2 mapping, T2* mapping and late gadolinium enhancement(LGE) sequences, as well as LVEF and extracellular volume(ECV) to evaluate the respective changes before and after anthracycline chemotherapy.

DETAILED DESCRIPTION:
Osteosarcoma is the most common primary malignant bone tumor in children and young adults and accounts for 5% of all pediatric malignancies. The long-standing chemotherapy regimen of doxorubicin and cisplatin with or without methotrexate remains a standard treatment of osteosarcoma.But anthracyclines such as doxorubicin have a notorious cardiotoxic side effect, which causes chemotherapy-related cardiac dysfunction(CTRCD). The American Society of Echocardiography (ASE) and the European Association of Cardiovascular Imaging (EACVI) defines it as a decrease in left ventricular ejection fraction (LVEF) of more than 10% to below the lower limit of normal, which is considered an LVEF of 53%, despite symptoms.

Cardiac magnetic resonance imaging is the gold standard for detection of ventricular volume and function. The parametric mapping techniques provide a non-invasive tool for quantifying tissue alterations in myocardial disease and is capable of in vivo tissue characterization.

In this study, the investigators used a contrast-enhanced (CE) cardiac magnetic resonance imaging(CMR), which included the measurement of T1 mapping, T2 mapping, T2* mapping and late gadolinium enhancement(LGE) sequences, as well as LVEF and extracellular volume(ECV) to evaluate the respective changes before and after anthracycline chemotherapy.

Study Population:

This prospective study was conducted at the Second Affiliated Hospital, School of Medicine, Zhejiang University. All chemotherapy naive patients whose biopsy results show high grade osteosarcoma were considered. Patients with underlying heart disease, severe hypertension, diabetes mellitus and previous history of gadolinium contrast agent allergy were excluded.Patients were treated with a standard chemotherapy protocol containing anthracyclines.

Study Protocol:

All patients underwent a contrast-enhanced (CE) cardiac magnetic resonance imaging(CMR), including measurement of LVEF, T1mapping, T2mapping, T2*mapping, ECV, LGE before starting chemotherapy (baseline), after neoadjuvant chemotherapy treatment, at the end of treatment (within 1 month), or whenever required by the clinical situation. These times points corresponded to scheduled oncological controls.

The CMR protocol included a standard segmented cine steady-state free-precession sequence, a T2 gradient spin-echo mapping sequence, a T2* gradient spin-echo mapping sequence, native and post-contrast T1 mapping sequences, and late gadolinium enhancement (LGE) sequence. The imaging parameters for the standard segmented cine steady-state free-precession sequence were as follows: field of view (FOV) 340 X340 mm², slice thickness 8 mm , repetition time (TR) 34.84ms, echo time (TE) 1.14ms, flip angle 67°, voxel size 1.8 X1.8 mm, and number of excitation. The imaging parameters for the T2-gradient-spin-echo mapping sequence were FOV 340X 340 mm², acquisition voxel size 1.8 X1.8 mm², slice thickness 8 mm, 8 echo times ranging from 6.7 to 53.6ms, and flip angle 70°. The T2* mapping sequence parameter were FOV 340X340 mm², acquisition voxel size 1.3X1.3mm², slice thickness 8mm, 8 echo times ranging from 2.22 to 17.48 (2.22,4.4,6.58,8.76,10.94,13.12,15.3,17.48), and flip angle 20°. The T1 mapping sequence (Modified Look-Locker Inversion recovery [MOLLI]) was acquired before and 10 min after contrast administration. All MOLLI sequences were based on a 5(3)3 scheme using a single shot steady-state free precession readout sequence (TR/TI/TE/flip angle 291.84ms/183ms/1.22ms/35°) with an in-plane acquisition resolution of 1.2 X1.2 mm² and an 8mm slice thickness. LGE imaging was performed 8 min after intravenous administration of 0.2mmol/kg gadopentetate dimeglumine contrast agent using a 3-dimensional inversion-recovery spoiled turbo field echo sequence (TR/TE/flip angle 813.6ms/1.09ms/40). Inversion time was adjusted before acquisition using a look-locker scout sequence with different inversion times to ensure proper nulling of the healthy myocardium signal.

The primary end point of the study was completion of chemotherapy with anthracycline drugs.

The secondary end point was cardiotoxicity. The time of occurrence of cardiotoxicity was recorded. Cardiotoxicity was defined as an LVEF reduction >10% from baseline, or LVEF <53%.

The following cardiac events were also considered as secondary end points: cardiac death, acute coronary syndromes, acute pulmonary edema, overt HF, and life-threatening arrhythmias.

ELIGIBILITY:
Inclusion Criteria:

* All chemotherapy naive patients whose biopsy results show high grade osteosarcoma undergoing an anthracycline agent as part of their chemotherapy regimen
* Informed consent has been signed

Exclusion Criteria:

* Strict contraindications to contrast-enhanced cardiac magnetic resonance imaging
* Underlying heart disease:myocardial infarction, heart failure, valvular disease or cardiomyopathy
* Acute or chronic kidney failure

Ages: 8 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All chemotherapy naive patients whose biopsy results show high grade osteosarcoma undergoing an anthracycline agent as part of their chemotherapy regimen without the underlying heart disease.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Completion of chemotherapy with anthracycline drugs | Through study completion, an average of 6 months.
  Chemotherapy regimen completed.

SECONDARY OUTCOMES:
Incidence of Cancer therapy-related cardiac dysfunction | From start of anthracycline therapy up to 6 months of anthracycline completion
  Cancer therapy-related cardiac dysfunction was defined as an LVEF reduction >10% from baseline, or LVEF <53%

OTHER OUTCOMES:
Changes of T1 mapping values | At timepoints 0 months, 2 months and 6 months (corresponding to the chemotherapy regimen controls)
  Change in T1 mapping values before and after anthracyclin chemotherapy
Changes of T2 mapping values | At timepoints 0 months, 2 months and 6 months (corresponding to the chemotherapy regimen controls)
  Change in T2 mapping values before and after anthracyclin chemotherapy
Changes of T2* mapping values | At timepoints 0 months, 2 months and 6 months (corresponding to the chemotherapy regimen controls)
  Change in T2* mapping values before and after anthracyclin chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2015 Jan;28(1):1-39.e14. doi: 10.1016/j.echo.2014.10.003. PMID 25559473
- [Background] Chen Y, Huang T, Shi W, Fang J, Deng H, Cui G. Potential targets for intervention against doxorubicin-induced cardiotoxicity based on genetic studies: a systematic review of the literature. J Mol Cell Cardiol. 2020 Jan;138:88-98. doi: 10.1016/j.yjmcc.2019.11.150. Epub 2019 Nov 18. PMID 31751567
- [Background] Li J, Chang HM, Banchs J, Araujo DM, Hassan SA, Wagar EA, Yeh ETH, Meng QH. Detection of subclinical cardiotoxicity in sarcoma patients receiving continuous doxorubicin infusion or pre-treatment with dexrazoxane before bolus doxorubicin. Cardiooncology. 2020 Jan 2;6:1. doi: 10.1186/s40959-019-0056-3. eCollection 2020. PMID 32154027
- [Background] Kopp LM, Womer RB, Schwartz CL, Ebb DH, Franco VI, Hall D, Barkauskas DA, Krailo MD, Grier HE, Meyers PA, Wexler LH, Marina NM, Janeway KA, Gorlick R, Bernstein ML, Lipshultz SE; Children's Oncology Group. Effects of dexrazoxane on doxorubicin-related cardiotoxicity and second malignant neoplasms in children with osteosarcoma: a report from the Children's Oncology Group. Cardiooncology. 2019 Oct 28;5:15. doi: 10.1186/s40959-019-0050-9. eCollection 2019. PMID 32154021
- [Background] Puntmann VO, Valbuena S, Hinojar R, Petersen SE, Greenwood JP, Kramer CM, Kwong RY, McCann GP, Berry C, Nagel E; SCMR Clinical Trial Writing Group. Society for Cardiovascular Magnetic Resonance (SCMR) expert consensus for CMR imaging endpoints in clinical research: part I - analytical validation and clinical qualification. J Cardiovasc Magn Reson. 2018 Sep 20;20(1):67. doi: 10.1186/s12968-018-0484-5. PMID 30231886
- [Background] Messroghli DR, Moon JC, Ferreira VM, Grosse-Wortmann L, He T, Kellman P, Mascherbauer J, Nezafat R, Salerno M, Schelbert EB, Taylor AJ, Thompson R, Ugander M, van Heeswijk RB, Friedrich MG. Clinical recommendations for cardiovascular magnetic resonance mapping of T1, T2, T2* and extracellular volume: A consensus statement by the Society for Cardiovascular Magnetic Resonance (SCMR) endorsed by the European Association for Cardiovascular Imaging (EACVI). J Cardiovasc Magn Reson. 2017 Oct 9;19(1):75. doi: 10.1186/s12968-017-0389-8. PMID 28992817
- [Background] Haaf P, Garg P, Messroghli DR, Broadbent DA, Greenwood JP, Plein S. Cardiac T1 Mapping and Extracellular Volume (ECV) in clinical practice: a comprehensive review. J Cardiovasc Magn Reson. 2016 Nov 30;18(1):89. doi: 10.1186/s12968-016-0308-4. PMID 27899132
- [Background] Haslbauer JD, Lindner S, Valbuena-Lopez S, Zainal H, Zhou H, D'Angelo T, Pathan F, Arendt CA, Bug G, Serve H, Vogl TJ, Zeiher AM, Carr-White G, Nagel E, Puntmann VO. CMR imaging biosignature of cardiac involvement due to cancer-related treatment by T1 and T2 mapping. Int J Cardiol. 2019 Jan 15;275:179-186. doi: 10.1016/j.ijcard.2018.10.023. Epub 2018 Oct 11. PMID 30360992
- [Background] Altaha MA, Nolan M, Marwick TH, Somerset E, Houbois C, Amir E, Yip P, Connelly KA, Michalowska M, Sussman MS, Wintersperger BJ, Thavendiranathan P. Can Quantitative CMR Tissue Characterization Adequately Identify Cardiotoxicity During Chemotherapy?: Impact of Temporal and Observer Variability. JACC Cardiovasc Imaging. 2020 Apr;13(4):951-962. doi: 10.1016/j.jcmg.2019.10.016. Epub 2019 Dec 18. PMID 31864977
- [Result] Whelan JS, Bielack SS, Marina N, Smeland S, Jovic G, Hook JM, Krailo M, Anninga J, Butterfass-Bahloul T, Bohling T, Calaminus G, Capra M, Deffenbaugh C, Dhooge C, Eriksson M, Flanagan AM, Gelderblom H, Goorin A, Gorlick R, Gosheger G, Grimer RJ, Hall KS, Helmke K, Hogendoorn PC, Jundt G, Kager L, Kuehne T, Lau CC, Letson GD, Meyer J, Meyers PA, Morris C, Mottl H, Nadel H, Nagarajan R, Randall RL, Schomberg P, Schwarz R, Teot LA, Sydes MR, Bernstein M; EURAMOS collaborators. EURAMOS-1, an international randomised study for osteosarcoma: results from pre-randomisation treatment. Ann Oncol. 2015 Feb;26(2):407-14. doi: 10.1093/annonc/mdu526. Epub 2014 Nov 24. PMID 25421877
- [Result] Demissei BG, Hubbard RA, Zhang L, Smith AM, Sheline K, McDonald C, Narayan V, Domchek SM, DeMichele A, Shah P, Clark AS, Fox K, Matro J, Bradbury AR, Knollman H, Getz KD, Armenian SH, Januzzi JL, Tang WHW, Liu P, Ky B. Changes in Cardiovascular Biomarkers With Breast Cancer Therapy and Associations With Cardiac Dysfunction. J Am Heart Assoc. 2020 Jan 21;9(2):e014708. doi: 10.1161/JAHA.119.014708. Epub 2020 Jan 21. PMID 31959034